CLINICAL TRIAL: NCT01072227
Title: Identification and Characterization of the Bacteria Causing Acute Otitis Media (AOM) Episodes in Young Children in Taiwan
Brief Title: Study to Identify and Characterize the Bacteria Causing Acute Otitis Media Episodes in Young Children in Taiwan
Status: Terminated | Type: Observational
Why Stopped: The study was terminated for logistic reasons
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113932
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Acute Otitis Media
Keywords: Non-typeable Haemophilus Influenzae; Acute Otitis Media; Streptococcus Pneumoniae; Etiology
MeSH Terms: conditions — Otitis Media | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue

GROUPS / COHORTS (1):
- Single Group
  Interventions: Procedure: Sample Collection

INTERVENTIONS:
Procedure: Sample Collection — Tissue

SUMMARY:
The purpose of the study is to identify the bacterial aetiology of Acute Otitis Media episodes in young children aged >= 3 months to < 5 years in Taiwan

ELIGIBILITY:
Inclusion Criteria:

* Age: >= 3 months and < 5 years at the time they are seen by the pediatrician or ear, nose and throat specialist. The subject becomes ineligible on the fifth birthday.
* Onset of signs and symptoms of acute otitis media within 72 hours:
* One of the functional or general signs of otalgia (, conjunctivitis, fever and either
* Paradise's criteria or
* Spontaneous otorrhea of less than 1 day.
* Written informed consent obtained from parent or legally acceptable representative prior to study start.

Exclusion Criteria:

* Hospitalized during the diagnosis of acute otitis media.
* Onset of otorrhea greater than 1 day prior to enrolment.
* Otitis externa, or otitis media with effusion.
* Presence of a transtympanic aerator.
* Systemic antibiotic treatment received for a disease other than acute otitis media in the 72 hours prior to enrolment.
* Receiving antimicrobial prophylaxis for recurrent acute otitis media.
* Provision of prescribing antibiotics by ear, nose and throat specialist and Pediatricians for acute otitis media before sample collection.
* Intended or planned prescription of antibiotic by pediatrician or ear, nose and throat specialist prior to the completion of study specified procedures during the enrolment visit.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects aged >= 3 months and < 5 years of age, diagnosed as having AOM in hospital by pediatricians or ear nose and throat (ENT) specialists.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Proportion of H. influenzae, S. pneumoniae and other bacterial pathogens | Average duration: 12 months

SECONDARY OUTCOMES:
Distribution of H. influenzae and S. pneumoniae serotypes. | Average duration: 12 months
Antimicrobial susceptibility of H. influenzae, S. pneumoniae and Moraxella catarrhalis | Average duration: 12 months
Proportion of treatment failure of Acute Otitis Media (AOM) and of recurrent AOM | Average duration: 12 months
Occurrence of spontaneous otorrhea | Average duration: 12 months
Occurrence of H. influenzae in AOM cases with treatment failure and in new AOM cases without treatment therapy | Average duration: 12 months
Occurrence of H. influenzae in AOM cases vaccinated with a pneumococcal vaccine. | Average duration: 12 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Taiwan (2):
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan Hsien